CLINICAL TRIAL: NCT05214404
Title: Effect and Mechanism of Dopamine on Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: Dopamine-UC
Record Dates: First submitted 2022-01-05; First posted 2022-01-28 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Dopamine Dysregulation Syndrome; Ulcerative Colitis
Keywords: Dopamine; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endoscopic biopsy specimens of colorectal mucosa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ulcerative colitis group: Patients with ulcerative colitis as observation group
  Interventions: Other: Patients diagnosed with ulcerative colitis
- Non-ulcerative colitis group: Non-ulcerative colitis as control group

INTERVENTIONS:
Other: Patients diagnosed with ulcerative colitis — Patients with ulcerative colitis diagnosed by endoscopy and histopathology
  Groups: Ulcerative colitis group

SUMMARY:
Increased evidence suggests that dopamine acts as an important regulator of immune function. A substantial amount of dopamine exists in the gastrointestinal tract, especially in colonic lumen. Decreased dopamine level has been reported in the colonic mucosa of ulcerative colitis patients. Therefore, the investigators suppose that colonic dopamine could involve in the ulcerative colitis and play an important role. This study aims to explore the role of dopamine in ulcerative colitis and underlying mechanism, which will provide a rationale for diagnosis and treatment of the ulcerative colitis.

DETAILED DESCRIPTION:
This study is a case-control clinical study. 30 patients with non-ulcerative colitis examined by endoscopy were selected as the control group. According to the inclusion and exclusion criteria, 30 patients with ulcerative colitis were determined. The baseline data of patients were recorded objectively: name, sex, age, vital signs, body weight and stool condition (frequency, character, etc.). Some laboratory examination results (blood routine, fecal routine and fecal culture, liver function, blood coagulation function, electrolyte, etc.), ulcerative colitis lesion range, ulcerative colitis classification and related history (common disease, treatment history and life history). Colonic mucosal tissue samples of patients with ulcerative colitis and control group were obtained by colonoscopic biopsy. The degree of inflammation was evaluated by related inflammatory factors via ELISA. The changes of dopamine system was detected by HPLC-ECD, Western Blot and immunohistochemistry. This study aims to provide new diagnostic and therapeutic basis, select appropriate drug delivery through clarify the effect and mechanism of local dopamine on colitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with or without ulcerative colitis diagnosed by endoscopy and histopathology
2. Negative bacterial culture in stool
3. Written informed consent

Exclusion Criteria:

1. Patients with cardiovascular and cerebrovascular diseases, or patients with severe impairment of liver, kidney and hematopoietic system
2. Mental patients
3. Hemorrhagic diseases
4. Platelet count < 50 × 10 ^ 9 / L
5. Allergic constitution
6. unable to tolerate or cooperate with endoscopy
7. Patients with serious complications, such as intestinal obstruction, intestinal perforation, toxic colonic dilatation, colorectal cancer, etc.
8. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with oulcerative colitis diagnosed by endoscopy and histopathology
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Comparison of the levels of inflammatory factors in colonic mucosa | 1 day
  The levels of inflammatory factors in colonic mucosa of ulcerative colitis group and non-ulcerative colitis control group were detected by Elisa to evaluate the degree of inflammation.
Comparison of dopamine content in colonic mucosa | 1 day
  HPLC-ECD was used to detect and compare the content of dopamine in colonic mucosa between ulcerative colitis group and non-ulcerative colitis group.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, MD, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of Chinese PLA General Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No